CLINICAL TRIAL: NCT03640117
Title: The Value of Geriatric Assessments in Predicting Treatment Tolerance and Overall Survival in Older Patients With Breast Cancer.
Brief Title: The Value of Geriatric Assessments in Older Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGAprediting
Record Dates: First submitted 2018-07-26; First posted 2018-08-21 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Aging; Breast Cancer; Chemotherapeutic Toxicity; Survival
Keywords: aging; geriatric assessment; chemotherapy toxicity; overall survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elderly cancer patients are a special group, often complicated by a variety of chronic diseases, which bring serious obstacles to surgery and adjuvant treatment. It is for these reasons that most patients with high-level evidence-based randomized controlled clinical trials will be part of these patients. Exclusions ultimately lead to a lack of standards for the treatment of elderly breast cancer patients, especially the chemotherapy.

Investigators' purpose was to determine whether geriatric assessments are associated with completion of a chemotherapy course, grade III/IV toxicity or survival in older adults with breast cancer in older patients.

Investigators want to prospectively enroll breast cancer patients with age ≥70 years. By recording the pre-treatment baseline laboratory tests and geriatric assessments, through questionnaires, including Karnofsky performance status(KPS), Eastern Cooperative Oncology Group(ECOG), Mini Nutritional Assessment(MNA), Activity of daily living(ADL), Instrumental activities of daily living(IADL), Mini-Mental State Examination(MMSE), Geriatric Depression Scale(GDS), G-8, Vulnerable Elders Survey-13（VES-13） and FRAIL, Tilburg. Investigators want to learn the relationship between the geriatric assessments and chemotherapy toxicity, chemotherapy completion and overall survival. Establish a model for predicting chemotherapy side effects in old breast cancer patients.

DETAILED DESCRIPTION:
Elderly cancer patients are a special group, often complicated by a variety of chronic diseases, which bring serious obstacles to surgery and adjuvant treatment. It is for these reasons that most patients with high-level evidence-based randomized controlled clinical trials will be part of these patients. Exclusions ultimately lead to a lack of standards for the treatment of elderly breast cancer patients, especially the chemotherapy. Numerous studies have shown that older adults are undertreated. This may be, in part, due to concerns about a greater risk of treatment toxicity in older adults.

Investigators' purpose was to determine whether geriatric assessments are associated with completion of a grade III/IV toxicity or survival in older adults with breast cancer in older patients. A predictive model that incorporates geriatric and oncologic correlates of vulnerability to chemotherapy toxicity in older adults could help both the healthcare provider and the patient weigh the benefits and risks of chemotherapy treatment and could serve as a platform to test interventions to decrease the risk of chemotherapy toxicity.

Investigators enroll the breast cancer patients ≥70y，the general data such as age, BMI, hemoglobin, white blood cells, creatinine, albumin, lactate dehydrogenase, blood pressure (diastolic blood pressure) were recorded; comorbidity scores using Charlson's Co-morbidity index（CCI） scores; a wide variety of comprehensive assessment scales for the elderly, after searching previous research and considering the operability of the actual data collected, the KPS, ECOG, MNA, ADL, IADL, MMSE, GDS, G-8, Vulnerable Elders Survey-13（VES-13） and FRAIL, Tilburg assessments were included. The treatment for these participants were decided by their own doctors. The participants who underwent chemotherapy were recorded for their chemotherapy regimen and dosage, and the side effects of chemotherapy were evaluated at the first cycle and after the end of the drug. The surgical methods, pathology after operation, radiotherapy and endocrine therapy also recorded. Long-term follow-up, record the participant's recurrence and recurrence time, cause of death and time. Investigators want to learn the relationship between the geriatric assessments and chemotherapy toxicity, chemotherapy completion and overall survival. Establish a model for predicting chemotherapy side effects in old breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed by pathology for breast cancer
* Patients aged 70 years and older

Exclusion Criteria:

* Patients with severe mental decline who cannot cooperate with the questionnaire

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In this prospective cohort study, patients aged 70 years and older with breast cancer, completed geriatric assessment questionnaire prior to therapy. For patients accepted chemotherapy, toxicity after chemotherapy were recorded using WHO criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of chemotherapy side effects using WHO criteria | two evaluations completed up to 6 months
  evaluation of chemotherapy side effects using WHO criteria after first circle of chemotherapy and the end of all the chemotherapy.The most serious one from the two evaluation will be used for data analysis to study the relationship between geriatric assessment and chemotherapy toxicity.

SECONDARY OUTCOMES:
overall-survival | 5 years
  the time from the date of the initial geriatric assessment until death, censored at the last clinical contact. the relationship between geriatric assessment and overall-survival.

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China